CLINICAL TRIAL: NCT00598403
Title: Multicentre, Prospective, Comparative, Randomized, Double-blind, Double-dummy Study to Assess the Efficacy and Safety of Cefditoren Pivoxil vs. Ciprofloxacin in Uncomplicated Acute Cystitis
Brief Title: Efficacy and Safety of Cefditoren Pivoxil Versus Ciprofloxacin in Acute Uncomplicated Cystitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tedec-Meiji Farma, S.A. (Industry)
Responsible Party: Mercedes Gimeno/ R&D Director, Tedec-Meiji Farma, S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TM-ME1207/311; 2007-001486-15
Record Dates: First submitted 2008-01-09; First posted 2008-01-21 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Urinary Tract Infections
Keywords: Cystitis
MeSH Terms: conditions — Urinary Tract Infections; Cystitis | interventions — cefditoren pivoxil; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cefditoren pivoxil
  Interventions: Drug: cefditoren pivoxil
- 2 (Active Comparator): Ciprofloxacin
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: cefditoren pivoxil — 400 mg, oral, single dose during 3 days
  Other Names: Meiact, Spectracef, Telo
  Arms: 1
Drug: Ciprofloxacin — 250 mg, oral, twice a day for 3 days
  Other Names: Ciprofloxacino Mabo
  Arms: 2

SUMMARY:
The main objective of the study is to comparatively assess the efficacy and tolerability of the drugs under study in the treatment of acute uncomplicated cystitis.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) are one of the most frequent reasons of surgery visits in Primary Care. More than 95 percent of UTIs are monomicrobial, although the microorganisms implied are varied, and the range of effective drugs could be extensive. The species most frequently isolated is Escherichia coli, with prevalence ranking between 85 and 90 percent of documented cases. E. coli has developed resistance to different antibiotics. Cefditoren is situated as a good candidate for the treatment of uncomplicated UTIs due to its spectrum of activity against E. coli. The study has been designed in accordance with the guidelines and recommendations in force to assess the efficacy of cefditoren pivoxil against ciprofloxacin, a drug which despite the increasing rate of resistance in some countries, continues to be a drug of choice for the treatment of uncomplicated UTIs.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adult females (>= 18)
* Clinical signs and symptoms of uncomplicated acute cystitis (dysuria, urgency, frequency, suprapubic pain) with symptoms starting <=72 hours prior the study entry
* Positive pre-treatment clean-catch midstream urine culture (>= 103 CFU/ml) and pyuria (10 leukocytes/mm3 or more than 5 leukocytes/field 40x magnification) within the 48 hours prior to inclusion in the study
* In vitro susceptibility testing of the isolated uropathogen to the drugs under study
* Written informed consent

Exclusion Criteria:

* Males
* Woman who are pregnant, nursing or not using a medically accepted, effective method of birth control
* Three or more episodes of uncomplicated acute infections of the urinary tract during the past 12 months
* Symptoms starting >4 days prior to admission
* Body temperature >= 38.3ºC, back pain, chills or other manifestations suggestive of upper urinary infection
* Evidence of structural or functional alterations of the urinary tract, such as calculi, stenosis, primary renal disease (eg. polycystic renal disease) or neurogenic bladder
* Underlying disease predisposing to complicated urinary tract infections such as diabetes mellitus, immunosuppression, leucopenia, heart insufficiency, liver impairment and neoplastic processes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Microbiological efficacy | 5-9 days post-therapy

SECONDARY OUTCOMES:
Clinical efficacy | 5-9 days post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Ballve, Principal Investigator; Josep R Toll, Principal Investigator; Rosa Viñas, Principal Investigator; Rosaura Figueras, Principal Investigator; Joan Palou, Principal Investigator; Gabriel Martín, Principal Investigator; Ramon Pons, Principal Investigator; Manel Terns, Principal Investigator; Josep L Fernandez, Principal Investigator; Pere Toran, Principal Investigator; Pilar Montero, Principal Investigator; Bingen Uriondo, Principal Investigator; Pablo Daza, Principal Investigator; Jesus Zorita, Principal Investigator; Ander Larrazabal, Principal Investigator; Natividad Gonzalez, Principal Investigator; Jose F Magdalena, Principal Investigator; Fernando Martin, Principal Investigator; Jose Porta, Principal Investigator; Mª Rosa Magallon, Principal Investigator; Mª Sol Reixa, Principal Investigator; Jesus Torrecilla, Principal Investigator; Isabel Blasco, Principal Investigator; Antonio Hidalgo, Principal Investigator; Alicia Alvarez, Principal Investigator; Gabriel Romera, Principal Investigator; Estrella Castro, Principal Investigator; Manuel M Ortega, Principal Investigator; Salvador Pertusa, Principal Investigator; Manuel Ramirez, Principal Investigator; Aggelos Pefanis, Principal Investigator; Chatzimouratidis, Principal Investigator; Jose V Vaquer, Principal Investigator; Nicolas Salvador, Principal Investigator; Jose L Pardo, Principal Investigator; Joaquin Aracil, Principal Investigator; Mª Jesus Barreda, Principal Investigator; Artemio Alvarez, Principal Investigator; Vicente Lopez, Principal Investigator; Panagiotis Gargalianos, Principal Investigator; Dolores M Maestre, Principal Investigator
Locations (30):
- Greece (2):
  - General Hospital of Chest Disease of Athens, Athens
  - General Hospital of Thessaloniki, Thessaloniki
- Spain (28):
  - CS Rincón de Loix, Benidorm, Alicante
  - CAP Cornella, Cornellà de Llobregat, Barcelona
  - CAP 17 setembre, el Prat de Llobregat, Barcelona
  - CAP Bartomeu Fabres Anglada, Gavà, Barcelona
  - CAP Amadeu Torner, L'Hospitalet de Llobregat, Barcelona
  - CAP Florida Nord, L'Hospitalet de Llobregat, Barcelona
  - CAP Dr. Vicens Papaceit, La Roca del Vallès, Barcelona
  - CAP Les Bases-Manresa 3, Manresa, Barcelona
  - CAP La Riera, Mataró, Barcelona
  - CAP El Maresme, Mataró, Barcelona
  - CAP Navas-Balsareny, Navàs, Barcelona
  - CAP Remei, Vic, Barcelona
  - CS San Telmo, Jerez de la Frontera, Cadiz
  - CS Cabra, Cabra, Cordoba
  - CS Lucena, Lucena, Cordoba
  - CS Rute, Rute, Cordoba
  - CS Billabona, Billabona, Guipuzcoa
  - CS Legazpi, Legazpi, Guipuzcoa
  - CS Monzón Urbano, Monzón, Huesca
  - CS Basurto, Bilbao, Vizcaya
  - CS Cabo Huertas, Alicante
  - CAP El Clot, Barcelona
  - Fundacion Puigvert, Barcelona
  - CS Sagasta Ruiseñores, Zaragoza
  - CS Torrero La Paz, Zaragoza
  - CS Torre Ramona, Zaragoza
  - CS Arrabal, Zaragoza
  - CS Bombarda, Zaragoza